CLINICAL TRIAL: NCT05679661
Title: Effect of Perioperative Immunonutrition Intervention and Oral Decontamination on Postoperative Complications in Elderly: a Prospective Randomized Controlled Trial
Brief Title: Perioperative Immunonutrition Intervention and Oral Decontamination in Elderly Surgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huang YuGuang (Other)
Responsible Party: Sponsor-Investigator, Huang YuGuang, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: K2870
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (immunonutrition and oral chlorhexidine decontamination, IN&CD) (Experimental): Patients will receive immunonutrition supplement of ORAL IMPACT™ 2 servings per day from the day of allocation at the preoperative anesthesia clinic until the day before surgery and oral chlorhexidine decontamination using 0.12% chlorhexidine oral rinse twice daily from the day before surgery until postoperative day 3.
  Interventions: Dietary Supplement: immunonutrition; Behavioral: oral chlorhexidine decontamination
- Group B (immunonutrition and routine oral care, IN&RC) (Experimental): Patients will receive immunonutrition supplement of ORAL IMPACT™ 2 servings per day from the day of allocation at the preoperative anesthesia clinic until the day before surgery and routine oral care.
  Interventions: Dietary Supplement: immunonutrition
- Group C (routine nutrition advice and oral chlorhexidine decontamination, RN&CD) (Experimental): Patients will be advised to follow a standard nutrition advice with a total intake of 30kcal/kg/d and protein intake of 1.2g/kg/d. Patients will also receive oral chlorhexidine decontamination using 0.12% chlorhexidine oral rinse twice daily from the day before surgery until postoperative day 3.
  Interventions: Behavioral: oral chlorhexidine decontamination
- Group D (routine nutrition advice and routine oral care, RN&RC) (No Intervention): Patients will be advised to follow a standard nutrition advice and routine oral care.

INTERVENTIONS:
Dietary Supplement: immunonutrition — Patients in the intervention group will receive additional immunonutrition supplementation, which is oral intake of ORAL IMPACT™ 2 servings per day from the day of allocation at the preoperative anesthesia clinic until the day before surgery.
  Arms: Group A (immunonutrition and oral chlorhexidine decontamination, IN&CD); Group B (immunonutrition and routine oral care, IN&RC)
Behavioral: oral chlorhexidine decontamination — Patients in the intervention group will receive oral chlorhexidine decontamination using 0.12% chlorhexidine oral rinse twice daily from the day before surgery until postoperative day 3.
  Arms: Group A (immunonutrition and oral chlorhexidine decontamination, IN&CD); Group C (routine nutrition advice and oral chlorhexidine decontamination, RN&CD)

SUMMARY:
Elderly patients are vulnerable to postoperative complications. Preoperative malnutrition and poor oral hygiene are risk factors for postoperative complications especially pulmonary complications. This study aims to investigate the feasibility and efficacy of perioperative oral decontamination and immunonutrition supplement on reducing postoperative complications in elderly surgical patients.

DETAILED DESCRIPTION:
This study is a prospective, single center, two-by-two factorial randomized controlled trial to evaluate the feasibility and efficacy of perioperative oral chlorhexidine decontamination and immunonutrition supplementation on postoperative complications in elderly surgical patients. Patients aged 65 years and older who are scheduled for elective non-cardiac surgeries will be recruited and randomized into four groups in 1:1:1:1 ratio (oral decontamination vs routine oral care with/without immunonutrition supplementation).

ELIGIBILITY:
Inclusion Criteria:

1. age≥65 years;
2. undergoing non-cardiac surgery (expected duration >2 hours);
3. scheduled for general anesthesia and endotracheal intubation;
4. ASA classification I-IV;
5. with intermediate to high risk of respiratory complications assessed by ARISCAT score (Assess Respiratory Risk in Surgical Patients in Catalonia);
6. inform consent obtained

Exclusion Criteria:

1. emergency surgery;
2. preoperative pneumonia;
3. allergic to chlorhexidine;
4. severe hepatic/renal dysfunction, incapable of oral feeding, with autoimmune diseases, taking immunosuppressant or immunoregulation medications, or with other contraindication to immunonutrition supplementation;
5. expected intervention of immunonutrition<3 days.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | within 7 days after surgery
  evaluated by trained investigator

SECONDARY OUTCOMES:
postoperative pneumonia | within 7 days after surgery
  defined according to the US Centers for Disease Control Definition
postoperative recovery | within 30 days after surgery
  evaluated by QoR-15 and WHODAS2.0
Comprehensive complication index (CCI) | within 30 days after surgery
  postoperative complication evaluated using Comprehensive complication index
Length of hospital stay | From date of surgery until discharge day, assessed up to 4 weeks
  Postoperative length of hospital stay assessed by days

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, Principal Investigator — Peking Union Medical College Hospital (CAMS)
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No